CLINICAL TRIAL: NCT06306898
Title: Intra-Arrest-Ventilation - a Prospective Randomized Trial in Human Cadavers
Brief Title: Intra-Arrest-Ventilation in Human Cadavers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerrit Jansen (Other)
Collaborators: Ruhr University of Bochum (Other); Bielefeld University (Other)
Responsible Party: Sponsor-Investigator, Gerrit Jansen, Principal Investigator, Muehlenkreiskliniken, MKK
Organization: Muehlenkreiskliniken, MKK (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IAV-2024-01
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Arrest
Keywords: ventilation; airway management
MeSH Terms: conditions — Heart Arrest; Respiratory Aspiration | interventions — Intubation, Intratracheal; Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: Randomized crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IPPV (Active Comparator): Intermittend-Positive-Pressure-Ventilation
  Interventions: Other: Endotracheal Intubation; Other: Laryngeal tube; Other: Laryngeal mask; Other: I-Gel-Laryngeal Mask
- CCSV (Active Comparator): Chest Compression Synchronized Ventilation
  Interventions: Other: Endotracheal Intubation; Other: Laryngeal tube; Other: Laryngeal mask; Other: I-Gel-Laryngeal Mask
- Bag-Device-Ventilation (Active Comparator): Ventilation with a Ventilation Bag
  Interventions: Other: Endotracheal Intubation; Other: Laryngeal tube; Other: Laryngeal mask; Other: I-Gel-Laryngeal Mask

INTERVENTIONS:
Other: Endotracheal Intubation — Ventilation with an endotracheal tube
Other: Laryngeal tube — Ventilation with an laryngeal tube
Other: Laryngeal mask — Ventilation with an laryngeal mask
Other: I-Gel-Laryngeal Mask — Ventilation with an I-Gel-laryngeal mask

SUMMARY:
The study investigates the influence of non-synchronized bag-device-ventilation and intermittent positive pressure ventilation (IPPV), as recommended in the current resuscitation guidelines of the European Resuscitation Concil (tidal Volume (Vt) = 5-6 mL/kg body weight, respiratory rate = 10 min-1) and Chest Compression Synchronized Ventilation (pInsp = 40 mbar; respiratory rate = chest compression rate) with regard to achieving a sufficient tidal volume and the tightness of various supraglottic airway devices (laryngeal mask, i-Gel-laryngeal mask, laryngeal tube) and endotracheal intubation.

DETAILED DESCRIPTION:
The European Resuscitation Council (ERC) guidelines for cardiopulmonary resuscitation (CPR) recommend uninterrupted chest compressions and continuous ventilation as soon as a patient is endotracheally intubated or a supraglottic airway (SGA) is positioned.

Recently, SGAs have been adopted by emergency medical services worldwide as the primary tool for airway management during CPR. SGAs offer limited protection against aspiration compared to endotracheal intubation (ETI) and may increase the risk of aspiration. A new ventilation mode (Chest Compression Synchronized Ventilation [CCSV]) is now available for resuscitation with uninterrupted chest compressions.

The study investigates the influence of non-synchronized bag-device-ventilation, intermittent positive pressure ventilation (IPPV), as recommended in the current resuscitation guidelines of the ERC (Vt = 5-6 mL/kg bw, AF = 10 min-1) and CCSV (pInsp = 40 mbar; RR = chest compression rate) with regard to achieving a sufficient tidal volume and the tightness of various SGA (laryngeal mask, iGel, laryngeal tube) and endotracheal intubation.

Gender, age, height and weight are documented (external post-mortem examination). The respective body donor is randomly assigned to a group. The grouping determines the order in which the means of airway management (SGA, ETI) are used.

Initial airway management is performed with an ETI with blockage of 30 mmH2O). The body donor is then bronchoscoped. A gastric tube is placed and the pressure probe to be used is calibrated if necessary. Positive pressure ventilation (pInsp = 40 mbar, positive end-expiratory pressure (PEEP) = 12 mbar, frequency = 10 min-1) is performed for 2 minutes to recruit the lungs. Vt is documented.

Mechanical cardiopulmonary resuscitation (CPR) is then performed for minutes (4 cycles) using the mechanical chest compression device in accordance with ERC 2015. Ventilation pressure and flow curves are continuously recorded by the respirator (Medumat Standard², Weinmann GmbH). Leaks are detected via the automatically initiated ventilation curves, measured and recorded by the ventilator. Ventilation takes place for 4 minutes with bad-device-ventilation, 4 minutes in IPPV mode and 4 minutes in CCSV mode. At the end of the two cycles, the body donor is intubated with one of the remaining airway devices, and the lungs are recruited again and mechanical CPR is performed again for 12 minutes using the 3 ventilation modes.

ELIGIBILITY:
Inclusion Criteria:

* > 17 Years of Age

Exclusion Criteria:

* Adult respiratory distress syndrome (ARDS)
* Severe lung or thoracic injuries
* pneumothorax
* Abnormal airways
* Tracheostoma
* severe aspirations

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Expiratory Volume with different Airway Devices in IPPV | After beginning of ventilation up to 4 minutes each device
  Mean expiratory Volume with different Airway Devices in IPPV
Ventilation Pressure with different Airway devices in CCSV | After beginning of ventilation up to 4 minutes each device

CONTACTS AND LOCATIONS:
Locations (1):
- JWK Minden, Minden, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lohmann J, Brand-Saberi B, Ullrich M, Gelashvili T, Hoyer A, Kolaparambil Varghese LJ, Kuehn V, Neuhaus C, Schneider C, Trenkel J, Hinkelbein J, Jansen G. Influence of different airway devices on intra-arrest ventilation during bag-valve-device ventilation - a prospective randomized controlled cadaver study. Crit Care. 2025 Dec 5;29(1):519. doi: 10.1186/s13054-025-05713-z. PMID 41345669
- [Derived] Gelashvili T, Brand-Saberi B, Darvishali M, Hoyer A, Kolaparambil Varghese LJ, Kuehn V, Lohmann J, Neuhaus C, Schneider C, Trenkel J, Hinkelbein J, Jansen G. Efficacy of supraglottic airway devices in chest compression synchronized ventilation during continuous resuscitation: a prospective randomized cross-over cadaver study. Resuscitation. 2025 Nov;216:110795. doi: 10.1016/j.resuscitation.2025.110795. Epub 2025 Sep 2. PMID 40907692